CLINICAL TRIAL: NCT04636034
Title: The Effect of Ganglion Sphenopalatine Block (SPG-block) Versus Placebo on Persistent Headache Following COVID-19 Infection: a Randomised, Blinded, Clinical Trial
Brief Title: The Effect of Ganglion Sphenopalatine Block Versus Placebo on Persistent Headache Following COVID-19 Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mads Seit Jespersen, MD, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSPB-COVID-2020
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Headache; Covid19; Sphenopalatine Ganglion Block; Persistent Headache Following COVID-19
MeSH Terms: conditions — Headache; COVID-19 | interventions — Sphenopalatine Ganglion Block; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ropivacaine-Lidocaine (Experimental)
  Interventions: Procedure: Sphenopalatine Ganglion Block with Local Anesthetic
- Placebo (Placebo Comparator)
  Interventions: Procedure: Sphenopalatine Ganglion Block with Placebo (Isotone NaCl)
- "Sham"-block with Placebo (Sham Comparator)
  Interventions: Procedure: "Sham"-block with Placebo (Isotone NaCl)

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block with Local Anesthetic — Block performed with bilaterally inserted q-tips with 1:1 mixture of lidocaine 40mg/ml and ropivacaine 5mg/mL
  Arms: Ropivacaine-Lidocaine
Procedure: Sphenopalatine Ganglion Block with Placebo (Isotone NaCl) — Block performed with bilaterally inserted q-tips with isotone NaCl
  Arms: Placebo
Procedure: "Sham"-block with Placebo (Isotone NaCl) — Block performed with bilaterally inserted q-tips with isotone NaCl. The q-tips are inserted a maximum of 3 cm into the nasopharynx thus not reaching the mucus above the ganglion.
  Arms: "Sham"-block with Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of the ganglion sphenopalatine block (SPG block) on persistent headache following acute COVID-19 infection.

DETAILED DESCRIPTION:
Adult patients with persistent headache following COVID-19 infection will be enrolled in the study. The patients will be randomised into three groups; bilateral SPG-block withto receive local anesthetic (lidocaine + ropivacaine), bilateral SPG-block with placebo (isotone NaCl) or bilateral "sham"-block with placebo (isotone NaCl).

Primary outcome is hyperactivity in the sphenopalatine ganglion assessed by pain intensity (0-100mm on a visual analogue scale, VAS) of the headache in standing position 30 minutes after block in the group Ropicavain-Lidocain and "sham".

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Moderate to severe headache (NRS >= 3) with self reported duration of minimum 6 hours during the past week as well as moderate to severe headache (NRS >= 3) on the day of intervention.
* Onset of headache during or maximum 4 weeks after PCR-verified COVID-19 infection.
* Headache must have persisted for at least 4 weeks following COVID-19 diagnosis.

Exclusion Criteria:

* Patients who cannot cooperate to the study
* Patients who does not understand or speak Danish
* Allergy to the drugs used in the study
* Has taken opioids within 12 hours prior to intervention
* History of migraine or persistent headache before COVID-19 infection.
* Active COVID-19 infection (defined by the Danish Goverment regulations, i.e. 48 hours after last symptoms (omitting long term effects) or 7 days after positive COVID-19 test if no symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Hyperactivity in the sphenopalatine ganglion assessed by pain intensity (0-100mm on a visual analogue scale, VAS) of the postdural headache in standing position in the group Ropivacine-Lidocaine and "sham". | 30 minutes after block
  Pain intensity will be measured as worst experienced pain after the patient has been standing for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.

SECONDARY OUTCOMES:
Number of patients with pain rating below 30mm in standing position (0-100mm on a visual analogue scale, VAS) | 30 minutes and 1 week after block
  Pain intensity measured as worst experienced pain after the patient has been standing for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.
Worst experienced pain in standing position (0-10 on a numercial rating scale, NRS) | During study period until completion of 1 week follow up
  The worst experienced pain reported during the week following the block as registered by the patient.
Average pain intensity (0-10 on a numercial rating scale, NRS) | During study period until completion of 1 week follow up
  The average pain intensity reported during the week following the block as registered by the patient.
Number of patients needing "rescue GSP-block" | At 1 week follow up
  If the patient at the 1 week follow up still needs further treatment a "rescue SPG-block" defined as a new SPG-block with "open label" analgetics will be offered.
Hyperactivity in the sphenopalatine ganglion assessed by pain intensity (0-100mm on a visual analogue scale, VAS) of the postdural headache in standing position in all 3 groups. | 30 minutes after block
  Pain intensity will be measured as worst experienced pain after the patient has been standing for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.

OTHER OUTCOMES:
Analgesics used daily in the week following the SPG-block | During study period until completion of 1 week follow up
  The use of analgesics during the week following the block as registered by the patient and the patient file.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, PhD, Study Director — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg and Frederiksberg Hospital, University of Copenhagen, Copenhagen, Denmark